CLINICAL TRIAL: NCT00791622
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study Evaluating QT/QTc Intervals Following Administration of Extended-release Paliperidone and Quetiapine in Subjects With Schizophrenia or Schizoaffective Disorder
Brief Title: A Study of QT and QTc Intervals in Patients Administered Extended Release Paliperidone or Quetiapine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR011056
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Paliperidone ER; Schizophernia; Mood Disorders, Antipsychotic drugs; Cardiovascular; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mood Disorders | interventions — Paliperidone Palmitate

INTERVENTIONS:
Drug: Paliperidone ER

SUMMARY:
The purpose of this study is to 1) determine whether the effect on QT interval corrected (QTcLD) for heart rate using the population specified linear derived method at steady state is comparable between 12 mg paliperidone extended-release (ER) once daily and that of 400-mg quetiapine administered twice daily, 2) to explore the relationship between the pharmacokinetics of paliperidone ER and electrocardiogram (ECG) parameters of interest, 3) to explore the cardiovascular safety and tolerability of 18 mg paliperidone ER at steady state, and 4) to evaluate the safety and tolerability of all treatments.

DETAILED DESCRIPTION:
This multicenter, placebo- and positive-controlled, randomized study consists of 3 phases - a screening phase of up to 5 days, a 6-day placebo washout phase, and a treatment phase that includes 1-day of open-label moxifloxacin treatment (Day 1), 10 days of double-blind treatment (Days 2 to 11), and end of study evaluations (Day 12). On Day 1, all patients will receive open-label treatment with a single dose of 400 mg moxifloxacin administered in the morning. Moxifloxacin will be used to establish assay sensitivity on the QTc interval. Patients will then be randomly assigned to receive double-blind treatment with placebo, paliperidone ER, or quetiapine on Days 2 to 11. Two doses of paliperidone ER will be studied: 12 mg/day that is the maximum recommended dose and 18 mg/day that is a supratherapeutic dose (50% above the maximum recommended). Patients randomly assigned to paliperidone ER will be administered 12 mg on Days 2 to 6, 15 mg on Day 7, and 18 mg on Days 8 to 11. Patients randomly assigned to quetiapine will receive 100 mg bid on Day 2, 200 mg twice daily (bid) on Day 3, 300 mg bid on Day 4, and 400 mg bid on Days 5 to 11. Patients will receive double-blind study drug 30 minutes after having a standardized breakfast on Days 2 to 11. Serial time matched 12 lead ECG triplicate readings will be recorded on Days -2, -1, 6, and 11 (predose and 1, 1.5, 2.5, 3.5, 4.5, 6, and 12 hours postdose) as well as Day 1 (predose, 1, 1.5, 2.5, 3.5 hours postdose) and Days 7 and 12 (23.5 hours postdose). This study will explore the QTc and pharmacokinetic data from paliperidone ER (commercial formulation) and quetiapine (marketed atypical antipsychotic of the same therapeutic class) at the maximum recommended doses for both products and at a supratherapeutic dose (50% above the maximum proposed labeled dose) for paliperidone ER. Safety and tolerability will be monitored throughout the study.

A single oral dose of moxifloxacin 400 mg tablet on Day 1; Oral paliperidone ER 12 mg on Days 2 to 6; 15 mg on Day 7, and 18 mg on Days 8 to 11; Oral quetiapine 100 mg twice daily (bid) on Day 2; 200 mg bid on Day 3; 300 mg bid on Day 4; and 400 mg bid on Days 5 to 11.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder as defined by DSM-IV-TR criteria, with stable symptoms. Symptom stability is based on the clinical judgment of the investigator but should include as a minimum: no exacerbation of psychotic symptoms or psychiatric hospitalization for at least 3 months before screening and a CGI-S score of < =4 (moderate) at screening and Day -1
* Must have a normal 12-lead ECG at screening and on Days -1 and -2, including: Normal sinus rhythm (heart rate between 50 and 100 beats per minute
* QTcB interval < = 430 milliseconds for men, < = 450 milliseconds for women
* QRS interval < 110 milliseconds
* PR interval < 200 milliseconds
* Must weigh > = 50 kg ( > = 110 lb), with a BMI > = 18 and < = 35 kg/m2
* If female, must be postmenopausal for at least 2 years, surgically sterile, abstinent, or agree to practice an effective method of birth control if they are sexually active before entry and throughout the study. Effective methods of birth control include: abstinence, prescription oral contraceptives, contraceptive injections, intrauterine device, double barrier method, contraceptive patch, and male partner sterilization. Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at baseline before receiving a dose of study drug

Exclusion Criteria:

* Meets DSM-IV criteria for substance dependence in the 3 months before screening
* Is at risk for suicidal or violent behavior, as judged by the investigator
* Has a clinically significant abnormality on ECG at screening or on Days 2 and -1 of the study
* Has a heart rhythm disturbance that is known or suggested by history or that is demonstrated on ECG at screening, or on Days -2 and -1 of the study
* Has a blood pressure outside of the normal range (supine systolic blood pressure < 90 or > 140 mmHg or diastolic blood pressure < 60 or > 90 mmHg)
* Has unusual T-wave morphology in a majority of leads of the ECG (such as bifid T waves, low T waves) or prominent U waves at screening
* Has a history of additional risk factors for torsade de pointes, such as heart failure, hypokalemia, family history of known short or long QT syndrome, or sudden unexplained death at a young age (< = 40 years) in a first-degree relative (i.e., biological parent, sibling, or offspring)
* Has a relevant history of any significant and/or unstable cardiovascular, respiratory (including bronchial asthma), neurologic (including seizures or significant cerebrovascular disease), renal, hepatic, endocrine, immunologic, ophthalmologic, hematologic, or other systemic disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2006-01; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To determine whether the effect on QTcLD is comparable between 12-mg paliperidone ER at steady state and that of 400-mg quetiapine at steady state with twice daily dose administration.

SECONDARY OUTCOMES:
To explore the relationship between the pharmacokinetics of paliperidone ER and ECG parameters of interest, to evaluate the cardiovascular safety and tolerability of 18-mg paliperidone ER at steady state, and to evaluate overall safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of QT and QTc intervals in patients administered extended release paliperidone or quetiapine — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=725&filename=CR011056_CSR.pdf